CLINICAL TRIAL: NCT00731991
Title: The Effects of Active Release Technique and Proprioceptive Neurological Facilitation on Surface EMGs of Hypertonic Upper Trapezius Musculature
Brief Title: Art and Surface Electromyography (EMG)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Dr. James George, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR0408080128
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2008-08

CONDITIONS: Fatigue
Keywords: Muscle
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ART (Active Comparator): ART to the levator scapulae.
  Interventions: Other: ART
- PNF (Active Comparator): PNF to the levator scapulae.
  Interventions: Other: PNF
- Control (Placebo Comparator): No treatment will be given. The participant will sit in the treatment room with the doctor for 4 minutes.
  Interventions: Other: No Treatment

INTERVENTIONS:
Other: ART — ART to the levator scapulae.
  Arms: ART
Other: PNF — PNF to the levator scapulae.
  Arms: PNF
Other: No Treatment — No treatment will be given. The participant will sit in the treatment room with the doctor for 4 minutes.
  Arms: Control

SUMMARY:
The general purpose of this research project is to use surface electromyography to compare the effect of Active Release Technique versus Proprioceptive Neuromuscular Facilitation on the electrical activity of the upper trapezius muscle at rest and during contraction.

DETAILED DESCRIPTION:
Both ART and PNF are soft tissue techniques used to decrease muscle hypertonicity, myospasm, and/or trigger points and increase the overall function of muscles.

Active-release technique, or ART®, is a form of myofascial therapy used in pain management that involves soft-tissue manipulation. ART has the expressed goal of restoring optimal texture, motion, and function of the soft tissue while releasing entrapped nerves or blood vessels. An injury to a soft-tissue structure commonly causes the muscle to shorten to guard or protect the area. A clinician who is performing ART makes a soft contact with one hand on the patient just distal to the injured area while the other hand develops tension on the soft tissue. While the contact tension is maintained, the structure is lengthened using an "active motion." During the motion, the lesion is palpated and the physical contact with the patient is changed or moved slightly in order to concentrate the tension in the appropriate tissue (Swann, et al).

Active Release Technique was developed by Dr. Michael Leahy and is widely used in rehabilitative and sports medicine for myofacial pain syndromes. The ART group will be treated by one investigator in concurrence with treatment methods outlined in Dr. Leahy's ART instructional manual. An ART treatment pass involves taking the tissue from a shortened position to a lengthened position while the administer maintains manual contact. We will perform three passes of ART with a 10 second rest period between passes. We will only perform ART on the symptomatic side (side that fits inclusion criteria); if both sides are involved, each side will be considered as a separate analysis.

The research backing ART is inadequate. Although there are numerous testimonials, limited published research studies could be found. Dr. George's study of the effect of ART, HVLA and no treatment on the temporomandibular joint and masticatory muscles showed no significant difference between the pre- and post-treatment mouth opening measurements. Another ART study of lateral epicondylitis concluded that the technique was successful in removing adhesions and promoting restoration of normal tissue but also stated that research was inadequate (Howitt, et al). A carpal tunnel study completed in 2006 used EMG to measure the effectiveness of ART. There were significant improvement in symptom severity and functional status after treatment, but no significant differences found in the EMG analyses (George, Tepe, and Busold 119-122).

Proprioceptive neuromuscular facilitation (PNF) stretching techniques are commonly used in the athletic and clinical environments to enhance both active and passive range of motion (ROM) with a view to optimizing motor performance and rehabilitation by elongating the muscle (Sharman, et al).

A second investigator will perform all the PNF using the published protocol from Warren Hammer, DC, MS, DABCO, in the text Functional Soft Tissue Examination and Treatment by Manual Methods, which is as follows:

The patient is supine with the examiner supporting the head so that the neck is in contralateral sidebending and ipsilateral rotation and flexion. The whole cervical spine and occiput is fixed and held in long-axis traction. With the other hand, the examiner contacts the shoulder with the forearm parallel to the table and pushes inferiorly to determine end feel. While maintaining the above position, the examiner asks the patient to resist by pushing the shoulder superiorly against the examiner's resistance for 7 seconds. The examiner then asks the patient to let go and, while stabilizing the head and neck, depresses the shoulder as far as possible for 12 seconds.

A previous study of PNF concluded that the technique caused short-term deficits in strength, power output, and muscle activation; it also increased ranges of motion (Marek, et al). A second previous study concluded that PNF caused an increase in electromyographic activity of the masticatory muscles (Olivo, et al).

Surface EMG is a reliable, non-invasive tool used for measuring muscular electrical activity. Electromyography (EMG) can provide unique information about the mechanical and motor control strategies during various types of muscle actions. EMG measures muscle activation, with surface EMG reflecting the algebraic sum of electric muscle action potentials that pass within the recording areas of the EMG electrodes. There, EMG amplitude quantifies muscle activation, which can be altered by the number of motor units recruited and the firing rates of the activated motor units. Thus, decreases in EMG amplitude due to decreases in muscle activation (Marek, et al). The surface EMG protocol will be performed completely by a third investigator.

Farina, et al published an article showing that the EMG can give reliable indications of muscle activity and fatigue. A previous study of muscle activity using surface EMG noted that based on visual inspections, all surface EMG variables showed consistent linear to moderately curvilinear behavior as a function of time (Muhammed, et al). Surface EMG has been widely used and accepted however care must be taken in pad placement as incorrect placement will give readings of improper musculature, as concluded in a study by Susan Mercer.

ELIGIBILITY:
Inclusion Criteria:

* Not all of the below listed criteria must be present, but some combination of two or more should be present before the participant can be deemed to have hypertonic
* hypertonic levator scapulae musculature.
* Anterior head carriage
* Internally rolled shoulders
* Occupational risk of poor upper cross posture
* Palpable muscular tightness
* Tenderness to palpation of the area
* Participant complaint of pain or tightness in the area

Exclusion Criteria:

* Participants will be excluded from this study if they have a history of a trauma that lead to marked scar tissue in the upper trapezius muscle as this would alter the surface EMG readings due to injured and altered tissue.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Surface EMG | Participant receive Surface EMG then treatment with either ART or PNF followed by Surface EMG

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States